CLINICAL TRIAL: NCT05327842
Title: Evaluation of a Flexible Videoscope Training Simulator: a Randomized, Controlled, Simulation Teaching Study
Brief Title: Evaluation of a Flexible Videoscope Training Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wenlong Yao (101480), Associate Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TJMZK220405
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Difficult Airway
Keywords: intubation; flexible bronchoscope; difficult airway

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New training simulator (Experimental): Participants received training with new simulator
  Interventions: Device: New training simulator
- Traditional method (Active Comparator): Participants received traditional training
  Interventions: Device: Traditional simulator

INTERVENTIONS:
Device: New training simulator — Participants receive training with new simulator
  Arms: New training simulator
Device: Traditional simulator — Participants receive traditional training
  Arms: Traditional method

SUMMARY:
Flexible bronchoscope or videoscope plays important roles in managing difficult airway. But this technique is time-consuming and very difficult to learn for novices. The investigators design a simple training simulator to help them master this technique.

DETAILED DESCRIPTION:
In this study, residents without operational experience will be recruited. The training effect of the new simulator will be evaluated by comparison with traditional simulation teaching. Participants will receive training with the new simulator or traditional method for 1hour, and then they perform intubation with flexible videoscope in a simulated difficult airway model. The insertion time and success rate will be recorded. Last, they will complete the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Resident or Medical student
* Willing to participate to the study
* Consent to evaluate the measured data

Exclusion Criteria:

* experienced anesthetists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
insertion time | 1 hour
  time when participants perform flexible videoscope from incisor to carina

SECONDARY OUTCOMES:
success rate | 1 hour
  the rate of participants used flexible videoscope to view carina successfully

OTHER OUTCOMES:
Questionnaire | 1 hour
  A questionnaire was used to measure the self-evaluation of the trained persons

CONTACTS AND LOCATIONS:
Overall Officials: Wenlong Yao, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Z, Zhang K, Zhao X, Hu Y, He Y, Wan L, Yao W. Evaluation of a 12-hole clock model for improving bronchoscopic skills in simulated normal and difficult airways among anesthesia residents: A randomized controlled study. Medicine (Baltimore). 2024 Jun 7;103(23):e38510. doi: 10.1097/MD.0000000000038510. PMID 38847658